CLINICAL TRIAL: NCT01189110
Title: Auriculotherapy for Smoking Cessation
Brief Title: Auriculotherapy for Smoking Cessation: Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NRI 08-371
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2013-08

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; veterans; auriculotherapy
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Stimulation of auriculotherapy points on both ears with functioning Stim Flex 400A TENS unit once a week for 5 weeks.
  Interventions: Device: Auriculotherapy using TENS unit Stim Flex 400A
- Arm 2 (Placebo Comparator): Stimulation of auriculotherapy points on both ears with disabled Stim Flex 400A TENS unit once a week for 5 weeks.
  Interventions: Device: Auriculotherapy using TENS unit Stim Flex 400A

INTERVENTIONS:
Device: Auriculotherapy using TENS unit Stim Flex 400A — Although the mechanism of action of auriculotherapy is not well understood, the dominant scientific theory for how traditional acupuncture procedures works has suggested possible neurophysiologic and neurochemical pathways that may explain its effectiveness for treating specific disorders

SUMMARY:
Thirty three percent of our veterans currently smoke. Encouraging smoking cessation continues to be a top priority for the Veteran's Administration as smoking is the single most important preventable risk factor for mortality and morbidity. This study attempts to determine whether auriculotherapy may be used as an effective alternative to usual pharmacological interventions currently offered. Identifying an efficacious alternative method to nicotine patch or bupropion would be highly beneficial to veterans who want to quit smoking. This clinical trial took place at the Veterans Administration Medical Center, in conjunction with the smoking cessation clinic. One hundred twenty five veterans, male and female, age 19 or older, who smoked a minimum of 10 cigarettes per day, were evaluated for enrollment and randomized to two groups- true auriculotherapy and sham auriculotherapy in this 6 week trial.

DETAILED DESCRIPTION:
Methods: This randomized, double-blind, placebo-controlled clinical trial of 125 veterans was conducted to determine whether aural electrical stimulation (auriculotherapy) with the Stim Flex 400A TENS unit once a week for 5 consecutive weeks is associated with a higher rate of smoking abstinence are than observed with sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Do not meet any exclusion criteria; age 19 and above.

Exclusion Criteria:

Veterans will be excluded from the study if they:

* have history or current evidence of pathological condition of the ear (e.g. infection, inflammation, or skin disruption of the auricle
* are known to be pregnant (positive urine pregnancy test)
* have an indwelling cardiac pacemaker or defibrillator
* are actively psychotic (as evidenced by delusions, hallucinations, or disorganization), have a severe cognitive impairment, or current significant substance abuse disorder that might prevent full participation in this study. Also excluded are those who score greater than 20 on the PHQ-9 screening tool for depression
* refuse to sign an informed consent form
* have been on bupropion and/or nicotine patch in the past one month or intend to start bupropion and/or nicotine patch in the next 6 weeks.
* Have a urine cotinine level less than 3.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Jean Fritz, PhD, Principal Investigator — St. Louis VA Medical Center John Cochran Division, St. Louis, MO
Locations (1):
- St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri, United States

REFERENCES:
- [Result] Fritz DJ, Carney RM, Steinmeyer B, Ditson G, Hill N, Zee-Cheng J. The efficacy of auriculotherapy for smoking cessation: a randomized, placebo-controlled trial. J Am Board Fam Med. 2013 Jan-Feb;26(1):61-70. doi: 10.3122/jabfm.2013.01.120157. PMID 23288282

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between August 2010 and January 2011 at the St. Louis VA. The inclusion criteria were age 19 years or older and currently smoking ≥10 cigarettes per day.
  Two hundred thirteen veterans who either responded to a mailing or were referred by their primary care physician expressed interest in the study.
Pre-assignment Details: Seventeen were excluded due to eligibility criteria. The remaining 196 were scheduled to attend a 1-hour smoking cessation class. Twenty-nine did not attend. Eleven did not keep the consent appointment. Another 31 did not enroll for other reasons. Thus, 125 participants were randomized: 64 to the intervention group and 61 to the placebo group.
Groups:
- Arm 1: Intervention- true Stim Flex treatment
- Arm 2: Placebo group- sham Stim Flex machine
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 64 (September, 2010) | 61
Completed | 64 (February, 2011) | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data, smoking history, fagerstrom nicotine dependence, stage of change, PHQ-9, Percieved stress scale, Minnesota withdrawal scale
Groups:
- Arm 1: Two separate Stim Flex machines will be used in this study: Machine A (usual care) will be a usual functioning machine which is FDA approved; Machine B (sham treatment) will be altered to disable the electrical current to flow to the probe. Otherwise both machines will be identical and function identical except at the time the electrical current is given thru the probe. There is no alteration to the outside of either Stem Flex machines, the alteration to the sham machine will be internal, and will appear and sound identical to the Stim Flex machine which has not been altered.
- Arm 2: Machine B (sham treatment) will be altered to disable the electrical current to flow to the probe. Otherwise both machines will be identical and function identical except at the time the electrical current is given thru the probe. There is no alteration to the outside of either Stem Flex machines, the alteration to the sham machine will be internal, and will appear and sound identical to the Stim Flex machine which has not been altered.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 61 | 125
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.1) | 55.8 (10) | 55.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 48 | 47 | 95
Region of Enrollment [Number; unit: participants]
  United States | 64 | 61 | 125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Self-reported Abstinence at 6 Weeks.
Description: Percentage of study participants free from smoking at 6 weeks based on self-report (yes/no).
Time Frame: 6 weeks
Population: A middle-aged, US military veteran population not free of smoking (at least 10 cigarettes per day) and not currently in reciept of any other form of smoking cessation intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm 1- Intervention: Receipt of auriculotherapy via a Stim Flex machine that provided full electrical flow of current to the ear probe.
- Arm 2- Placebo: Receipt of sham auriculotherapy via a Stim Flex machine that disabled electrical flow of current to the ear probe.
Arm/Group | Arm 1- Intervention | Arm 2- Placebo
Number analyzed (Participants) | 64 | 61
percentage of participants | 12.3 [4.0 to 20.7] | 12.9 [4.0 to 21.7]
Statistical Analysis 1: Comparison: Arm 1- Intervention vs Arm 2- Placebo; A two-proportion z-test was used to compare the proportion of self-reported abstinence at 3 weeks between groups; Test type: Superiority or Other; p = 0.74, Chi-squared; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.23 to 2.83], Standard Error of Mean 0.42

ADVERSE EVENTS:
Groups:
- Arm 1- Intervention: Two separate Stim Flex machines will be used in this study: Machine A (usual care) will be a usual functioning machine which is FDA approved; Machine B (sham treatment) will be altered to disable the electrical current to flow to the probe. Otherwise both machines will be identical and function identical except at the time the electrical current is given thru the probe. There is no alteration to the outside of either Stem Flex machines, the alteration to the sham machine will be internal, and will appear and sound identical to the Stim Flex machine which has not been altered.
- Arm 2- Placebo: Machine B (sham treatment) will be altered to disable the electrical current to flow to the probe. Otherwise both machines will be identical and function identical except at the time the electrical current is given thru the probe. There is no alteration to the outside of either Stem Flex machines, the alteration to the sham machine will be internal, and will appear and sound identical to the Stim Flex machine which has not been altered.
Arm/Group | Arm 1- Intervention | Arm 2- Placebo
Serious Adverse Events (participants affected / at risk) | 2/64 | 0/61
Other Adverse Events (participants affected / at risk) | 0/64 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- Intervention (N=64) | Arm 2- Placebo (N=61)
hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — one hospitalization for psychiatric reasons not related to study
hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
It is possible that the pressure alone applied to these points provided a therapeutic effect and therefore was not a true placebo.

Other stimulation frequencies or intensities may have produced a different outcome condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No